CLINICAL TRIAL: NCT02091973
Title: MicroRNA Expression in Everolimus-based Versus Tacrolimus-based Maintenance Immunosuppressive Regimens in Kidney Transplantation
Brief Title: MicroRNA Expression in Everolimus-based Versus Tacrolimus-based Regimens in Kidney Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wiwat Chancharoenthana, Dr., Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WWC-004
Record Dates: First submitted 2014-03-18; First posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: microRNA Profiles
Keywords: everolimus; tacrolimus; kidney transplantation; microRNA
MeSH Terms: interventions — Everolimus; Tacrolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus (Experimental): everolimus dosing to tough level 6-10 ng/ml
  Interventions: Drug: Everolimus
- Tacrolimus (Experimental): Tacrolimus dosing to target tough level 5-10 ng/ml
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus dosing to target tough level 6-10 mg/ml
  Arms: Everolimus
Drug: Tacrolimus — Tacrolimus dosing to target tough level 5-10 ng/ml
  Arms: Tacrolimus

SUMMARY:
The calcineurin inhibitor drugs including cyclosporin and tacrolimus are well-known as nephrotoxicity. However, these drugs are essential for kidney transplant especially in high immunological risks. To date, however, there is an alternative regimen by using of everolimus-based which showing less toxicity than tacrolimus-based regimen by its mechanisms. Of note, this study aims to evaluate the toxicity by using microRNA profiles detection between everolimus-based and tacrolimus-based immunosuppressive regimen in kidney transplantation.

DETAILED DESCRIPTION:
The author aims to evaluate the effects of two regimens (everolimus-based versus tacrolimus-based) in kidney transplantation recipients. Both of regimens are prescribed only in recipents who have low immunologicla risks. After informed consent, all eligible recipients will be collected blood and urine sample for microRNA profile testing during study periods.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given informed consent to participate in the study
* Actual eGFR > 20-25 ml/min/1.73 m2

Exclusion Criteria:

* Multi-organ transplantation
* Pregnancy
* ABO incompatible blood group
* Second, third, fouth kidney transplantation
* HIV positive, active or carrier in any infections

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
microRNA profiles | 5 years
  microRNA profiles including rejection and nephrotoxicity markers

SECONDARY OUTCOMES:
Allograft tissue pathology | At year 2 and 5
  Pathology studies including rejection, interstitial fibrosis and tubular atrophy

CONTACTS AND LOCATIONS:
Overall Officials: Wiwat Chancharoenthana, MD, Msc., Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Thailand